CLINICAL TRIAL: NCT01323803
Title: Eosinophilic Esophagitis (EoE) Databank (CoFAR 5)
Brief Title: Eosinophilic Esophagitis Databank
Acronym: CoFAR5
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT CoFAR5
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Esophagitis; Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis
MeSH Terms: conditions — Esophagitis; Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood and saliva
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will establish a registry for participants with eosinophilic esophagitis (EoE) and create a research resource that will provide further insights into EoE.

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EoE) is a newly recognized chronic disease that is increasingly being diagnosed in children and adults. Many patients with EoE also have food allergies. EoE is characterized by inflammation and accumulation of a specific type of immune cell, called an eosinophil, in the esophagus. While there have been several large studies of EoE, very few have focused on the roles the immune system, genetics/heredity, and the environment in EoE.

The samples and information collected from participants will help to identify and understand the genetic mechanisms underlying eosinophilic esophagitis.

The Cincinnati Children's Hospital Medical Center will serve as the Central Laboratory for genetic characterization studies.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent from participant and consent from parent/guardian for minors with agreement for genetic testing;
* Documented diagnosis of EoE at any time confirmed by study team (pathology report describing greater than or equal to 15 eosinophils/hpf in peak field of an esophageal biopsy. Participants with eosinophilia in extra-esophageal tissue are permitted).

Exclusion Criteria:

* Participants with known infectious causes of esophageal eosinophilia such as esophageal fungus, gastric H. pylori, or systemic parasites;
* Participants with a history of persistent eosinophilia greater than 1500 cells/mcl of blood.

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with biopsy proven Eosinophilic Esophagitis
Sampling Method: Probability Sample
Enrollment: 709 (Actual)
Dates: Start 2011-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Elucidate the genetic components of EoE, focusing on a candidate gene approach the TSLP/WDR36 locus and through GWAS analysis | 48 months
  A Genome-Wide Association Study (GWAS) analysis of single-nucleotide polymorphisms (SNPs) from >1.5 million genetic markers will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Marc E. Rothenberg, M.D., Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati; Mirna Chehade, MD, MPH, Principal Investigator — Mt. Sinai School of Medicine
Locations (5):
- United States (5):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - National Jewish Health, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina

REFERENCES:
- [Result] Kottyan LC, Davis BP, Sherrill JD, Liu K, Rochman M, Kaufman K, Weirauch MT, Vaughn S, Lazaro S, Rupert AM, Kohram M, Stucke EM, Kemme KA, Magnusen A, He H, Dexheimer P, Chehade M, Wood RA, Pesek RD, Vickery BP, Fleischer DM, Lindbad R, Sampson HA, Mukkada VA, Putnam PE, Abonia JP, Martin LJ, Harley JB, Rothenberg ME. Genome-wide association analysis of eosinophilic esophagitis provides insight into the tissue specificity of this allergic disease. Nat Genet. 2014 Aug;46(8):895-900. doi: 10.1038/ng.3033. Epub 2014 Jul 13. PMID 25017104
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) — https://www.niddk.nih.gov/